CLINICAL TRIAL: NCT05431764
Title: Whole-target Consolidation Therapy After Standard Chemotherapy for Initial Diagnosed Distant Metastatic Nasopharyngeal Carcinoma Under Full-course Immunotherapy: An Open-Label, Single Center, Nonrandomized, Phase 2 Study
Brief Title: Whole-target Consolidation Therapy Under Systemic Therapy for Oligometastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-SBRT2022
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Oligometastatic Nasopharyngeal Carcinoma; Immunotherapy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Cisplatin; Immune Checkpoint Inhibitors; Radiosurgery; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Plus Stereotactic Body Radiotherapy (Experimental): Patients were treated with gemcitabine, cisplatin and camrelizumab for 6 cycles, followed by whole-target radiotherapy (IMRT for locoregional lesion and SBRT for oligometastatic lesions) and camrelizumab maintenance therapy.
  Interventions: Drug: Camrelizumab, gemcitabin, cisplatin; Radiation: Stereotactic Body Radiotherapy, Intensity modulated-radiotherapy

INTERVENTIONS:
Drug: Camrelizumab, gemcitabin, cisplatin — Patients receive gemcitabine (1000 mg/m² d1,8), cisplatin (80mg/m² d1), and camrelizumab (200mg, iv drip for over 60min) every 3 weeks for 6 cycles before locoregional radiotherapy.
  Other Names: PD-1 inhibitor
Radiation: Stereotactic Body Radiotherapy, Intensity modulated-radiotherapy — IMRT: 5 fractions per week for 6 weeks to a total dose of 70 Gy and 33 fractions to the primary tumor.
  SBRT: 3 months after locoregional IMRT, patients receive SBRT for all oligometastatic lesions as radical therapy to control the disease and reduce any potential adverse impact to living quality. The dosage is based on published clinical studies.
  Camrelizumab (200mg, iv drip for over 60min) every 2 weeks began on the first day of IMRT until an intolerable toxicity, or disease progression, or withdrawal of consent, or the investigator determines that he or she has to withdraw from treatment, or has been treated for up to 2 years.
  Other Names: SBRT; IMRT

SUMMARY:
In this exploratory clinical trial, patients with newly diagnosed distant metastatic nasopharyngeal carcinoma were treated with gemcitabine+ cisplatin+PD-1 inhibitor regimen followed by whole-target radiotherapy (IMRT for local regional lesion, SBRT for distant metastasis) and PD-1 inhibitor long-term maintenance regimen. To investigate the efficacy and safety of "whole target" radiotherapy combined with immuno-maintenance therapy.

DETAILED DESCRIPTION:
This exploratory clinical trial will evaluate tumor control rate, survival, and safety of newly diagnosed distant metastatic nasopharyngeal carcinoma by further adding local regional IMRT, distant metastatic SBRT and immuno-maintenance therapy to the standard regimen of gemcitabine+ cisplatin+ PD-1 inhibitor (historical data). To explore whether the "full target" model can be a better comprehensive therapy for the initial diagnosed distant metastatic nasopharyngeal carcinoma in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age.
2. Had histopathologically confirmed nonkeratinizing metastatic NPC that was diagnosed as stage IVb NPC (AJCC, 8th; the metastatic tissue biopsy is preferred, not necessary).
3. Patients who had not received anti-tumor therapy for nasopharyngeal cancer before this clinical trial.
4. Patients evaluated to have a partial response (PR) or stable disease (SD) by head and neck MRI and PET/CT after 3 months of locoregional radiotherapy, and the metastatic lesions were assessed as oligometastatic lesions (the number of total metastatic lesions no more than 5 and the number of metastatic lesions within a single organ no more than 3).
5. Stereotactic body radiotherapy applicable for all metastatic lesions according to MDT.
6. ECOG performance status of 0 or 1.
7. Maximum diameter of brain metastatic lesion no more than 3cm.
8. Maximum diameter of metastatic lesion (brain excluded) no more than 5cm.

   * Maximum diameter of bone metastatic lesion no more than 6cm if attending doctor decides it is safe to apply the treatment.
9. Life expectancy more than 6 months.

Exclusion Criteria:

1. History of severe hypersensitivity to any ingredient of PD-1/PD-L1 or other monoclonal antibody.
2. chemotherapy (cytotoxic or molecular targeted) within 4 weeks before stereotactic body radiotherapy.
3. Imageological evidence for spinal cord compression, or tumor less than 3mm away from spinal cord.
4. Patient with brain metastasis who needs decompression surgery.
5. Other malignancy or malignant hydrothorax.
6. Concurrent known or suspicious autoimmune disease, including dementia and epilepsy.
7. CHD no less than grade 2, arrhythmia (QTc interval over 450ms for male and 470ms for female) or cardiac insufficiency.
8. Use of large dose corticosteroids within 4 weeks before study drug administration.
9. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids.
10. Active tuberculosis (TB), anti-TB treatment is ongoing or within 1 year prior to screening
11. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy.
12. Has a known history of human immunodeficiency virus (HIV), has hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
13. Received any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment.
14. Pregnancy or lactation.
15. Other ineligible patients according to attending doctor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | 2 years
  Progression-free survival is calculated from the date of randomization to the date of death of any cause or the first progress at any site, censored on the last date of tumor evaluation if no progress has happened.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Objective response rate is the rate of patients achieving complete response or partial response for a certain period of time after intervention.
Disease control rate (DCR) | 2 years
  Disease control rate is the rate of patients achieving complete response, partial response or stable disease for at least 4 weeks after intervention.
Median overall survival (OS) | 2 years
  Overall survival is calculated from the date of randomization to the date of death of any cause, censored on the last date of known survival if no death has happened
Adverse events | 2 years
  NCI-CTC5.0 and RTOG standards are adopted, and acute subjective toxicity, acute objective toxicity and late subjective toxicity are included.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, and after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.
Duration of response (DoR) | 2 years
  Defined as the time from first documentation of objective response to radiological disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China